CLINICAL TRIAL: NCT03084822
Title: Cardiovascular Health Promotion Among African-Americans by FAITH! (Fostering African-American Improvement in Total Health): Engaging the Community Through Mobile Technology-assisted Education
Brief Title: Cardiovascular Health Promotion Among African-Americans by FAITH!
Acronym: FAITH!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Mayo Clinic Clinic Center for Innovation (Unknown); Mayo Clinic Center for Clinical and Translational Science (CCaTS) (Unknown)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Assistant Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-000353
Record Dates: First submitted 2017-03-01; First posted 2017-03-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Prevention; Physical Activity; Diet Modification; Diabetes; Hypertension; High Cholesterol; Pre Diabetes; Smoking Cessation; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Glucose Intolerance; Smoking Cessation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAITH! App digital intervention (Experimental): The digital app will include 10 education modules addressing the major CVD risk factors to be delivered on-demand through an innovative, interactive video series. The digital app will also support the multi-media education modules, interactive surveys/quizzes, self-monitoring (diet, physical activity), and social networking (discussion board) functionality.
  Interventions: Behavioral: FAITH! App digital intervention

INTERVENTIONS:
Behavioral: FAITH! App digital intervention — The digital app will include 10 education modules addressing the major CVD risk factors to be delivered on-demand through an innovative, interactive video series. The digital app will also support the multi-media education modules, interactive surveys/quizzes, self-monitoring (diet, physical activity), and social networking (discussion board) functionality.

SUMMARY:
Given the importance of healthy lifestyle practices to cardiovascular disease (CVD) prevention and the utility of church-based interventions in African-American adults, the investigators developed a theory-informed, strategically-planned, health and wellness intervention with Rochester, Minnesota (MN) and Twin Cities area (Minneapolis, St. Paul, MN) churches with predominately African-American congregations. The objective of the study was to partner with churches to implement a multi-component, health education program through the use of core educational sessions delivered through a digital-application accessible on demand via interactive access on computer tablets and the Internet. The overarching goal was to increase the awareness and critical importance of healthy lifestyles for CVD prevention and provide support for behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Basic Internet navigation skills, at least weekly Internet access, active email address, minimal fruit/vegetable intake (<5 servings/day), no regular physical activity program (< 30 minutes/d of moderate physical activity), able to engage in moderate physical activity (no restrictions)

Exclusion Criteria:

* Diagnosis of a serious medical condition or disability that would make participation difficult (i.e. visual or hearing impairment, mental disability that would preclude independent use of the app)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Diet (fruit/vegetable intake using adaptation of NIH Eating at America's Table Quick Food Scan Screener) | 28 weeks post-intervention
  Change in self reported diet
Physical activity behavior | 28 weeks post-intervention
  Change in self-reported physical activity, reported as minutes per week of moderate to vigorous physical activity
Diet self-efficacy (using Self-Efficacy and Eating Habits Survey) | 28 weeks post-intervention
  Change from baseline self-efficacy; scale of 1-5; Healthy diet score components include the following: fruits and vegetables, ≥4.5 cups/d; fish, 2 or more 3.5-oz servings/wk; fiber-rich whole grains (≥1.1 g fiber/10 g carbohydrate), 3 or more 1-oz-equivalent servings/d; sodium, ≤1500 mg/d; and sugar-sweetened beverages, ≤450 kcal/wk. Dietary recommendations are scaled according to a 2000-kcal/d diet.
Physical activity self-efficacy (using Self-Efficacy and Exercise Habits Survey) | 28 weeks post-intervention
  Change from baseline self-efficacy. Physical activity is reported via the Self-Regulation Scale from Health Beliefs Survey, which includes 10 items, using a 5-point Likert scale (1=never to 5=always) with higher scores indicating higher PA self-regulation

SECONDARY OUTCOMES:
Intervention feasibility | 28 weeks post-intervention
  Participant retention (goal >80% of enrolled participants)
BMI | 28 weeks post-intervention
  Change from baseline BMI
Blood Pressure | 28 weeks post-intervention
  Change from baseline blood pressure
Fasting Cholesterol | 28 weeks post-intervention
  Change from baseline cholesterol
Fasting glucose | 28 weeks post-intervention
  Change from baseline fasting glucose
Smoking (using adaptation of Global Adult Tobacco Survey) | 28 weeks post-intervention
  Change in self reported smoking status
Life's Simple 7 Composite Score | 28 weeks post-intervention
  Change from baseline Life's Simple 7 Composite Score; calculated as a composite of each LS7 component by assigning 2 points for ideal, 1 point for intermediate, or 0 points for poor. The total composite score is assessed on a scale of 0 to 14 points. To categorize, scores of 0 to 6 were labeled "poor', 7 to 8 "intermediate" and 9 to 14 "ideal" cardiovascular health.
Cardiovascular health knowledge | 28 weeks post-intervention
  Change in percent correct from baseline knowledge and attitudes about CVD

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess C Brewer, MD, MPH, Principal Investigator — Mayo Clinic Department of Cardiovascular Medicine

REFERENCES:
- [Derived] Brewer LC, Kumbamu A, Smith C, Jenkins S, Jones C, Hayes SN, Burke L, Cooper LA, Patten CA. A Cardiovascular Health and Wellness Mobile Health Intervention Among Church-Going African Americans: Formative Evaluation of the FAITH! App. JMIR Form Res. 2020 Nov 17;4(11):e21450. doi: 10.2196/21450. PMID 33200999
- [Derived] Brewer LC, Hayes SN, Caron AR, Derby DA, Breutzman NS, Wicks A, Raman J, Smith CM, Schaepe KS, Sheets RE, Jenkins SM, Lackore KA, Johnson J, Jones C, Radecki Breitkopf C, Cooper LA, Patten CA. Promoting cardiovascular health and wellness among African-Americans: Community participatory approach to design an innovative mobile-health intervention. PLoS One. 2019 Aug 20;14(8):e0218724. doi: 10.1371/journal.pone.0218724. eCollection 2019. PMID 31430294